CLINICAL TRIAL: NCT02985398
Title: An Open Label Phase 3 Trial to Evaluate the Safety of ALD403 Administered Intravenously in Patients With Chronic Migraines
Brief Title: An Open Label Trial of ALD403 (Eptinezumab) in Chronic Migraine
Acronym: PREVAIL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alder Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ALD403-CLIN-013
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Results first posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Migraine Disorder
MeSH Terms: conditions — Migraine Disorders | interventions — eptinezumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ALD403 (Eptinezumab) Dose Level 1 (Experimental): ALD403 (Eptinezumab) Dose Level 1 (IV)
  Interventions: Biological: ALD403 (Eptinezumab)

INTERVENTIONS:
Biological: ALD403 (Eptinezumab)
  Other Names: Eptinezumab-jjmr; Vyepti

SUMMARY:
An evaluation of long term safety of repeat ALD403 doses in Chronic Migraine

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 65 years of age, inclusive, who were diagnosed with migraines at ≤ 50 years of age, and have a history of chronic migraine for ≥ 12 months before screening.

Exclusion Criteria:

* Receipt of any monoclonal antibody treatment (within or outside a clinical trial) within 6 months before screening.
* Confounding and clinically significant pain syndromes (e.g. fibromyalgia, chronic low back pain, complex regional pain syndrome).
* Psychiatric conditions that are uncontrolled and/or untreated, including conditions that are not controlled for a minimum of 6 months prior to screening. Patients with a lifetime history of psychosis, mania, or dementia are excluded.
* History or diagnosis of complicated migraine (ICHD-III beta version, 20134), chronic tension-type headache, hypnic headache, cluster headache, hemicrania continua, new daily persistent headache, or sporadic and familial hemiplegic migraine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Research Site, San Diego, California
  - Research Site, Santa Monica, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Bradenton, Florida
  - Research Site, DeLand, Florida
  - Massachusetts, Miami, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Haven, Florida
  - Research Site, Prairie Village, Kansas
  - Massachusetts, Boston, Massachusetts
  - Research Site, North Attleboro, Massachusetts
  - 02481, Wellesley, Massachusetts
  - Research Site, Minneapolis, Minnesota
  - Research Site, Brooklyn, New York
  - Research Site, Rochester, New York
  - Research Site, Dayton, Ohio
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Fort Worth, Texas
  - Research Site, Bellevue, Washington

REFERENCES:
- [Derived] Blumenfeld A, Ettrup A, Hirman J, Ebert B, Cady R. Long-term reductions in disease impact in patients with chronic migraine following preventive treatment with eptinezumab. BMC Neurol. 2022 Jul 8;22(1):251. doi: 10.1186/s12883-022-02774-3. PMID 35804294
- [Derived] Smith TR, Spierings ELH, Cady R, Hirman J, Schaeffler B, Shen V, Sperling B, Brevig T, Josiassen MK, Brunner E, Honeywell L, Mehta L. Safety and tolerability of eptinezumab in patients with migraine: a pooled analysis of 5 clinical trials. J Headache Pain. 2021 Mar 30;22(1):16. doi: 10.1186/s10194-021-01227-5. PMID 33781209
- [Derived] Kudrow D, Cady RK, Allan B, Pederson SM, Hirman J, Mehta LR, Schaeffler BA. Long-term safety and tolerability of eptinezumab in patients with chronic migraine: a 2-year, open-label, phase 3 trial. BMC Neurol. 2021 Mar 19;21(1):126. doi: 10.1186/s12883-021-02123-w. PMID 33740902

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 158 participants signed the ICF, of which 128 participants met the entry criteria and were randomized into the trial.
Groups:
- 300 mg ALD403: Participants were enrolled and scheduled to receive 4 ALD403 IV infusions on Day 0, 84 (Week 12), 168 (Week 24), and 252 (Week 36), then up to 4 additional infusions at Weeks 48, 60, 72 and 84.
Period: Overall Study
Arm/Group | 300 mg ALD403
Started | 128
Participants Treated | 128
Completed | 106
Not Completed | 22
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 8
Not completed — Study Burden | 9

BASELINE CHARACTERISTICS:
Population: Safety Population includes all participants who received study drug.
Groups:
- 300 mg ALD403: Participants were randomized to receive 4 ALD403 IV infusions on Day 0, 84 (Week 12), 168 (Week 24), and 252 (Week 36), then up to 4 additional infusions at Weeks 48, 60, 72 and 84.
Arm/Group | 300 mg ALD403
Number analyzed (Participants) | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (11.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26
  Not Hispanic or Latino | 102
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 122
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 128
Duration of migraine diagnosis at baseline [Mean (Standard Deviation); unit: years] | 21.2 (11.65)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment Emergent Adverse Events (TEAEs)
Description: Treatment emergent adverse events were defined as adverse events with start date and time on or after the date and time of the initial study drug infusion.
Time Frame: 104 Weeks
Population: Safety Population includes all participants who received study drug.
Measure: Count of Participants; unit: Participants
Groups:
- 300 mg ALD403: Participants received 4 ALD403 IV infusions on Day 0, 84 (Week 12), 168 (Week 24), and 252 (Week 36), then up to 4 additional infusions at Weeks 48, 60, 72 and 84.
Arm/Group | 300 mg ALD403
Number analyzed (Participants) | 128
Participants | 91

2. Primary Outcome: Number of Participants With a Clinically Significant Electrocardiogram
Description: Overall investigator interpretation of participant electrocardiogram
Time Frame: Baseline, Day 0 Postdose, Week 12, 24, 36, 48 60, 72 and 84 (Predose and Postdose), and Week 104
Population: Safety Population includes all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403
Number analyzed (Participants) | 128
Participants
  Baseline | 0
  Day 0 Postdose | 1
  Week 12 Predose | 0
  Week 12 Postdose | 0
  Week 24 Predose | 0
  Week 24 Postdose | 0
  Week 36 Predose | 0
  Week 36 Postdose | 0
  Week 48 Predose | 0
  Week 48 Postdose | 0
  Week 60 Predose | 1
  Week 60 Postdose | 1
  Week 72 Predose | 1
  Week 72 Postdose | 1
  Week 84 Predose | 1
  Week 84 Postdose | 0
  Week 104 | 1

3. Primary Outcome: Number of Participants With Any Clinically Significant Laboratory Values
Description: Each of the laboratory values that were reported as abnormal and clinically significant and entered as adverse events in the database.
Time Frame: 104 Weeks
Population: Safety Population includes all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403
Number analyzed (Participants) | 128
Participants
  Hematocrit Decreased | 1
  Hemoglobin Decreased | 1
  Blood Glucose Increased | 1
  Hypertriglyceridemia | 1
  Blood Potassium Decreased | 1
  Hypokalemia | 1
  Blood Mercury Abnormal | 1
  Hypercholesterolemia | 1
  Hyperlipidemia | 1

4. Primary Outcome: Number of Participants Experiencing Suicidal Ideation or Suicidal Behavior on Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: Baseline responses are collected at screening and assess suicidal ideation in the past 6 months. Post baseline reports the worst assessment of suicidal ideation since the last visit for all post baseline visits.
Time Frame: 104 Weeks
Population: Safety Population includes all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403
Number analyzed (Participants) | 128
Participants
  Participants Experiencing Suicidal Ideation | 0
  Participants Experiencing Suicidal Behavior | 0

5. Primary Outcome: Number of Participants With Any Clinically Significant (CS) Changes in Vital Signs
Description: Changes in vital signs that were considered clinically meaningful or clinically significant (CS) by the Investigator
Time Frame: 104 Weeks
Population: Safety Population includes all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403
Number analyzed (Participants) | 128
Participants
  Number of CS changes in diastolic blood pressure | 0
  Number of CS changes in systolic blood pressure | 0
  Number of CS changes in heart rate value | 0

6. Secondary Outcome: Patient Global Impression of Change (PGIC) at Week 104
Description: The PGIC includes a single question concerning the participant's impression of the change in their disease status since the start of the study. Seven responses are possible: Very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse.
Time Frame: Week 104
Population: Safety Population includes all participants who received study drug. Only participants who completed the Week 104 Visit are included
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403
Number analyzed (Participants) | 96
Participants
  Very Much Improved | 47
  Much Improved | 33
  Minimally Improved | 11
  No Change | 5
  Minimally Worse | 0
  Much Worse | 0
  Very Much Worse | 0

7. Secondary Outcome: Change in Baseline of Short Form Health Survey (SF-36 v 2.0) Scale Scores
Description: The SF-36 is a health survey consisting of 36 questions consisting of eight scaled scores to measure quality of life over the past 4 weeks (scale range: 0=worst to 100=best). Increases from baseline indicate improvement.
Time Frame: Baseline to Week 12
Population: Safety Population includes all participants who received study drug. Only participants who completed the Week 12 Visit are included
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 300 mg ALD403
Number analyzed (Participants) | 124
score on a scale
  Bodily Pain | 5.8 (10.06)
  General Health | 1.6 (6.46)
  Mental Component | 1.9 (7.89)
  Mental Health | 1.4 (7.86)
  Physical Component | 4.5 (7.08)
  Physical Functioning | 2.9 (6.15)
  Role Emotional | 2.3 (9.09)
  Role Physical | 4.8 (8.34)
  Social Functioning | 4.9 (9.13)
  Vitality | 3.0 (7.90)

8. Secondary Outcome: Health Related Quality of Life (EQ-5D-5L) at Week 12
Description: The EQ-5D-5L is a descriptive health-related quality of life states consisting of 5 dimensions/questions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of five responses. The responses record five levels of severity (no problems/slight problems/moderate problems/severe problems/extreme problems) within a particular EQ-5D dimension.
Time Frame: Week 12
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403
Number analyzed (Participants) | 124
Participants
  Mobility: No problems | 110
  Mobility: Slight problems | 11
  Mobility: Moderate problems | 3
  Mobility: Severe problems | 0
  Mobility: Extreme problems | 0
  Self-care: No problems | 121
  Self-care: Slight problems | 3
  Self-care: Moderate problems | 0
  Self-care: Severe problems | 0
  Self-care: Extreme problems | 0
  Usual Activities: No problems | 95
  Usual Activities: Slight problems | 18
  Usual Activities: Moderate problems | 11
  Usual Activities: Severe problems | 0
  Usual Activities: Extreme problems | 0
  Pain/Discomfort: No problems | 55
  Pain/Discomfort: Slight problems | 42
  Pain/Discomfort: Moderate problems | 22
  Pain/Discomfort: Severe problems | 5
  Pain/Discomfort: Extreme problems | 0
  Anxiety/Depression: No problems | 96
  Anxiety/Depression: Slight problems | 22
  Anxiety/Depression: Moderate problems | 6
  Anxiety/Depression: Severe problems | 0
  Anxiety/Depression: Extreme problems | 0

9. Secondary Outcome: Change in Baseline of Headache Impact Test (HIT-6) Score
Description: The HIT-6 measures the impact of headache on the participant's functional health and well-being in 6 domains: pain; role functioning (ability to carry out usual activities); social functioning; energy or fatigue; cognition; and emotional distress assess over the prior 12-week period. The total possible scores range from 36 (no impact) to 78 (worst impact). The change in baseline will be calculated from the average scores.
Time Frame: Baseline, Week 1-4, Week 9-12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 300 mg ALD403
Number analyzed (Participants) | 128
score on a scale
  Week 1-4: number analyzed (Participants) | 126
  Week 1-4 | -8.0 (8.06)
  Week 9-12: number analyzed (Participants) | 124
  Week 9-12 | -7.9 (7.96)

10. Secondary Outcome: Change in Most Bothersome Symptom at Week 48
Description: The Investigator verbally obtained the most bothersome symptom associated with the participant's migraine during the screening visit. The most bothersome symptom may include nausea, vomiting, sensitivity to light, sensitivity to sound, mental cloudiness, fatigue, pain with activity, mood changes, or other migraine related symptoms. Participants were asked to rate the improvement in this symptom from screening on a seven-point scale.
Time Frame: Baseline to Week 48
Population: Safety Population includes all participants who received study drug. Only participants who completed the Week 48 Visit are included
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403
Number analyzed (Participants) | 112
Participants
  Very Much Improved | 40
  Much Improved | 44
  Minimally Improved | 17
  No Change | 11
  Minimally Worse | 0
  Much Worse | 0
  Very Much Worse | 0

11. Secondary Outcome: Change From Baseline of Migraine Disability Assessment (MIDAS) Total Score
Description: The MIDAS questionnaire measures the effect headaches have on the participant's daily functioning. MIDAS is composed of five questions that ask about the participant's performance over the past 3 months. The response to each question is provided in number of days which are summed to determine the MIDAS total score and level of disability:
  0-5, MIDAS Grade I, little or no disability; 6-10, MIDAS Grade II, mild disability; 11-20, MIDAS Grade III, moderate disability; 21+, MIDAS Grade IV, severe disability;
  A higher value represents a worse outcome.
Time Frame: Baseline to Week 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 300 mg ALD403
Number analyzed (Participants) | 123
score on a scale | -36.3 (51.85)

12. Secondary Outcome: Development of Anti-ALD403 Antibody by Visit
Description: Serum blood samples were taken at visits to test for the development of antibodies to ALD403, or anti-drug antibodies (ADA). Participants who tested positive for anti-ALD403 antibodies at the time of the last study visit were asked to provide up to 2 additional blood samples for immunogenicity testing at approximately 3 month intervals for up to 6 months.
Time Frame: Baseline, Week 2, 4, 8, 12, 24, 36, 48, 72 and 104
Population: Safety Population includes all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403
Number analyzed (Participants) | 128
Participants
  Day 0: ADA Results: ADA Positive | 0
  Day 0: ADA Results: ADA Negative | 128
  Week 2 : ADA Results: number analyzed (Participants) | 127
  Week 2 : ADA Results: ADA Positive | 1
  Week 2 : ADA Results: ADA Negative | 126
  Week 4 : ADA Results: number analyzed (Participants) | 126
  Week 4 : ADA Results: ADA Positive | 0
  Week 4 : ADA Results: ADA Negative | 126
  Week 8 : ADA Results: number analyzed (Participants) | 125
  Week 8 : ADA Results: ADA Positive | 7
  Week 8 : ADA Results: ADA Negative | 118
  Week 12 : ADA Results: number analyzed (Participants) | 123
  Week 12 : ADA Results: ADA Positive | 11
  Week 12 : ADA Results: ADA Negative | 112
  Week 24 : ADA Results: number analyzed (Participants) | 120
  Week 24 : ADA Results: ADA Positive | 21
  Week 24 : ADA Results: ADA Negative | 99
  Week 36 : ADA Results: number analyzed (Participants) | 118
  Week 36 : ADA Results: ADA Positive | 9
  Week 36 : ADA Results: ADA Negative | 109
  Week 48 : ADA Results: number analyzed (Participants) | 113
  Week 48 : ADA Results: ADA Positive | 6
  Week 48 : ADA Results: ADA Negative | 107
  Week 72 : ADA Results: number analyzed (Participants) | 101
  Week 72 : ADA Results: ADA Positive | 4
  Week 72 : ADA Results: ADA Negative | 97
  Week 104 : ADA Results: number analyzed (Participants) | 96
  Week 104 : ADA Results: ADA Positive | 0
  Week 104 : ADA Results: ADA Negative | 96

13. Secondary Outcome: Summary of Neutralizing Properties of Anti-ALD403 Antibodies by Visit
Description: Any samples that were positive for anti-ALD403 antibody, there was additional testing to characterize the anti-ALD403 antibody for the potential to neutralize (NAb) ALD403 activity.
Time Frame: Baseline, Week 2, 4, 8, 12, 24, 36, 48, 72 and 104
Population: Safety Population includes all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg ALD403
Number analyzed (Participants) | 128
Participants
  Day 0: NAb Results: number analyzed (Participants) | 0
  Day 0: NAb Results: NAb Positive | 0
  Day 0: NAb Results: NAb Negative | 0
  Week 2 : NAb Results: number analyzed (Participants) | 1
  Week 2 : NAb Results: NAb Positive | 0
  Week 2 : NAb Results: NAb Negative | 1
  Week 4 : NAb Results: number analyzed (Participants) | 0
  Week 4 : NAb Results: NAb Positive | 0
  Week 4 : NAb Results: NAb Negative | 0
  Week 8 : NAb Results: number analyzed (Participants) | 7
  Week 8 : NAb Results: NAb Positive | 3
  Week 8 : NAb Results: NAb Negative | 4
  Week 12 : NAb Results: number analyzed (Participants) | 11
  Week 12 : NAb Results: NAb Positive | 8
  Week 12 : NAb Results: NAb Negative | 3
  Week 24 : NAb Results: number analyzed (Participants) | 21
  Week 24 : NAb Results: NAb Positive | 5
  Week 24 : NAb Results: NAb Negative | 16
  Week 36 : NAb Results: number analyzed (Participants) | 9
  Week 36 : NAb Results: NAb Positive | 1
  Week 36 : NAb Results: NAb Negative | 8
  Week 48 : NAb Results: number analyzed (Participants) | 6
  Week 48 : NAb Results: NAb Positive | 1
  Week 48 : NAb Results: NAb Negative | 5
  Week 72 : NAb Results: number analyzed (Participants) | 4
  Week 72 : NAb Results: NAb Positive | 0
  Week 72 : NAb Results: NAb Negative | 4
  Week 104 : NAb Results: number analyzed (Participants) | 0
  Week 104 : NAb Results: NAb Positive | 0
  Week 104 : NAb Results: NAb Negative | 0

ADVERSE EVENTS:
Time Frame: Baseline to Week 104 (end of study)
Arm/Group | 300 mg ALD403
All-Cause Mortality (participants affected / at risk) | 0/128
Serious Adverse Events (participants affected / at risk) | 5/128
Other Adverse Events (participants affected / at risk) | 49/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 300 mg ALD403 (N=128)
Anaphylactic Reaction (Immune system disorders) | 1
Pneumonia (Infections and infestations) | 1
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Conversion Disorder (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 300 mg ALD403 (N=128)
Bronchitis (Infections and infestations) | 7
Influenza (Infections and infestations) | 8
Nasopharyngitis (Infections and infestations) | 18
Sinusitis (Infections and infestations) | 10
Upper respiratory tract infection (Infections and infestations) | 10
Migraine (Nervous system disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-01-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT02985398/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/98/NCT02985398/SAP_001.pdf